CLINICAL TRIAL: NCT06794476
Title: Milieu Teaching-AV (MT-AV Pilot): a Pilot Study to Assess the Feasibility of an Adaptation of Milieu Teaching for Infant Siblings of Autistic Children That Encourages Looking to the Mouth
Brief Title: Milieu Teaching-AV (MT-AV Pilot)
Acronym: MT-AV Pilot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Jacob I. Feldman, Postdoctoral Fellow, Vanderbilt University Medical Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 150878; 1K99DC021501 (NIH)
Record Dates: First submitted 2024-12-26; First posted 2025-01-27 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-01

CONDITIONS: Autism Sibling; Autism Spectrum Disorder
Keywords: parent-mediated; caregiver-mediated
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: This study will utilize single-case research design studies, which are experimental and can be used to demonstrate the effects of treatment with as few as 1-3 participants. The investigators will specifically conduct up to two multiple probe across participants (MPP) design studies with caregiver/Baby Sib dyads. These studies will focus on whether caregivers can be trained to administer the proposed intervention and whether implementers (hereafter referred to as coaches) can conduct the sessions as manualized with a high degree of procedural fidelity. This experimental design also can be used to determine whether the pre-emptive intervention produces positive effects on the proximal child variable of looking to mouth of their caregiver. Each intervention session will be video recorded to have coders naïve to condition monitor the fidelity of procedures and caregiver strategy use.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be naive to the phase of treatment and the hypotheses. Additionally, there will be at least one naive member of the study team that can decide when to implement phase changes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Business as usual baseline (No Intervention): The first several sessions will be conducted in a business-as-usual baseline condition; these sessions will then be compared to the Milieu Teaching-AV condition. Entry into the Milieu Teaching-AV condition will be staggered across participants to ensure that observed changes are not due to other factors (e.g., history, maturation).
- Milieu Teaching-AV (Experimental): Following baseline sessions, there will be staggered entry into the experimental condition.
  Interventions: Behavioral: Milieu Teaching-AV

INTERVENTIONS:
Behavioral: Milieu Teaching-AV — In Milieu Teaching-AV, coaches will teach caregivers to engage the child in play or routines around a standardized set of toys, follow the child's attention or communication lead around these toys, and respond to the infant's communication acts by modeling and expanding those communication acts into more sophisticated strategies. While responding to infant communication acts, coaches will slowly move the referent of the infant's lead near the face at approximately the level of the mouth, wait for the infant to shift his/her gaze towards the new referent position if necessary, and provide all models, prompting, and expanding while maintaining placement of the referent near the mouth.
  Other Names: Enhanced Milieu Teaching; Prelinuistic Milieu Teaching
  Arms: Milieu Teaching-AV

SUMMARY:
This project will look at whether a novel approach to language intervention that encourages looking to audiovisual speech cues for infants with autistic older siblings (Baby Sibs), who are highly likely be diagnosed with autism or developmental language disorder (DLD). This study will specifically look at (a) whether caregivers find this approach to be easy to implement in their homes, (b) whether they find this approach to be acceptable, and (c) whether caregivers use the taught strategies in interactions with their infants.

DETAILED DESCRIPTION:
This project will test the feasibility and acceptability of a novel approach to language intervention based on Milieu Teaching (Milieu Teaching-AV) that encourages looking to audiovisual speech cues for infants with autistic older siblings (Sibs-autism), who are highly likely be diagnosed with autism or developmental language disorder (DLD). The main question[s] it aims to answer are:

1. Can caregivers be trained in Milieu Teaching-AV, such that they are using the trained strategies in play with their infant children?
2. Do caregivers find these procedures to be acceptable and feasible to use in their everyday life.

ELIGIBILITY:
Inclusion Criteria:

* an older sibling with an autism diagnosis, confirmed by either (a) a detailed developmental interview and administration of the Autism Diagnostic Observation Schedule or (b) by record review
* monolingual English-speaking household

Exclusion Criteria:

* adverse neurological history
* known genetic condition
* pre-term birth (gestation < 37 weeks)
* caregiver report of a diagnosed vision impairment or hearing loss

Ages: 5 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Caregiver strategy use | From enrollment to the end of the treatment (i.e., all baseline and treatment sessions, up to 20 weeks)
  Proportion of milieu teaching trials during a caregiver-child free play session wherein the caregiver moves the referent of the child's lead towards the mouth

SECONDARY OUTCOMES:
Caregiver attitudes on the feasibility of Milieu Teaching-AV - Quantitative | At the conclusion of the treatment (i.e., following all intervention sessions; up to 20 weeks)
  Caregiver attitudes towards the feasibility of this approach will be conducted via the Feasibility Intervention Measure Score (range of scores = 4-20)
Caregiver attitudes on the acceptability of Milieu Teaching-AV - Quantitative | At the conclusion of the treatment (i.e., following all intervention sessions; up to 20 weeks)
  Caregiver attitudes towards the feasibility of this approach will be conducted via the Acceptability of Intervention Measure Score (range of scores = 4-20)
Caregiver attitudes on the feasibility of Milieu Teaching-AV - Qualitative | At the conclusion of the treatment (i.e., following all intervention sessions; up to 20 weeks)
  Caregiver attitudes towards the feasibility of this approach will be conducted via the coding of a qualitative interview.
Caregiver attitudes on the acceptability of Milieu Teaching-AV - Qualitative | At the conclusion of the treatment (i.e., following all intervention sessions; up to 20 weeks)
  Caregiver attitudes towards the acceptability of this approach will be conducted via the coding of a qualitative interview.

OTHER OUTCOMES:
Infants' looking to the mouth of their caregiver | From enrollment to the end of the treatment (i.e., all baseline and treatment sessions, up to 20 weeks)
  The proportion of looks to the caregivers' mouth during a caregiver-child free play, as measured via eye tracking technology
Infants' looking to the mouth of a speaker | From enrollment to the end of the treatment (i.e., all baseline and treatment sessions, up to 20 weeks)
  The proportion of looks to the mouth of a speaking during a recorded monologue of infant-directed audiovisual speech in the infants' native speech as measured via eye tracking technology
Infants' vocabulary | End of the treatment (i.e., following all treatment sessions, up to 20 weeks)
  Infants' vocabulary will be measured the end of the study via the MacArthur-Bates Communicative Development Inventories: Words and Gestures checklist
Autism Diagnostic Observation Schedule (2nd edition) | 15 months of age
  The clinical best estimate of the infants' preliminary diagnostic outcome at final the timepoint will be obtained from the Autism Diagnostic Observation Schedule. This measure yields both a diagnostic category (i.e., Little-to-No Concern for Autism, Mild-to-Moderate Concern for Autism, and Moderate-to-Severe Concern for Autism) as well as a Social Affect score (range = 0-22) and a Restricted and Repetitive Behavior score (range = 0-8).
Caregiver-Child Engagement | From enrollment to the end of the treatment (i.e., all baseline and treatment sessions, up to 20 weeks)
  The proportion of intervals in which caregivers and infants engage in higher- and lower-order supported joint engagement
The Vineland Adaptive Behavior Scales | Enrollment and end of the treatment (i.e., following all treatment sessions, up to 20 weeks)
  One assessment utilized to measure infants' communication abilities will be the receptive and expressive communication age equivalency scores of the Vineland Adaptive Behavior Scales.
Mullen Scales of Early Learning | Enrollment and end of the treatment (i.e., following all treatment sessions, up to 20 weeks)
  One assessment utilized to measure infants' communication abilities will be the receptive and expressive language age equivalency scores of the Mullen Scales of Early Learning.
Communication and Symbolic Behavior Scales | Enrollment and end of the treatment (i.e., following all treatment sessions, up to 20 weeks)
  One assessment utilized to measure infants' communication abilities will be the Communication and Symbolic Behavior Scales. This measure will specifically be utilized to obtain an estimate of infant's consonant inventory (i.e., the number of consonant sounds infants use in canonical syllables during intentional communication acts)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Graphs with individual data points will be reported in manuscripts that share the primary study findings. Additionally, all data will be made available via an open repository (e.g., OSF, institutional repository) after publication.
Supporting Information: Study Protocol, SAP
Time Frame: IPD and supporting information will be made available following the publication of the study and will be available indefinitely.
Access Criteria: IPD for all continuously collected variables will be made available via graphs published in the manuscript. Following the publication of all primary analyses, data for all quantitative data will be posted on an institutional repository.

REFERENCES:
- [Background] Ledford JR, Barton EE, Severini KE, Zimmerman KN. A Primer on Single-Case Research Designs: Contemporary Use and Analysis. Am J Intellect Dev Disabil. 2019 Jan;124(1):35-56. doi: 10.1352/1944-7558-124.1.35. PMID 30715924
- [Background] Hampton LH, Rodriguez EM. Preemptive interventions for infants and toddlers with a high likelihood for autism: A systematic review and meta-analysis. Autism. 2022 Aug;26(6):1364-1378. doi: 10.1177/13623613211050433. Epub 2021 Oct 11. PMID 34628968
- [Background] Santapuram P, Feldman JI, Bowman SM, Raj S, Suzman E, Crowley S, Kim SY, Keceli-Kaysili B, Bottema-Beutel K, Lewkowicz DJ, Wallace MT, Woynaroski TG. Mechanisms by which Early Eye Gaze to the Mouth During Multisensory Speech Influences Expressive Communication Development in Infant Siblings of Children with and without Autism. Mind Brain Educ. 2022 Feb;16(1):62-74. doi: 10.1111/mbe.12310. Epub 2022 Jan 19. PMID 35273650
- [Background] Pons F, Bosch L, Lewkowicz DJ. Twelve-month-old infants' attention to the eyes of a talking face is associated with communication and social skills. Infant Behav Dev. 2019 Feb;54:80-84. doi: 10.1016/j.infbeh.2018.12.003. Epub 2019 Jan 8. PMID 30634137
- [Background] Tenenbaum EJ, Amso D, Abar B, Sheinkopf SJ. Attention and word learning in autistic, language delayed and typically developing children. Front Psychol. 2014 May 26;5:490. doi: 10.3389/fpsyg.2014.00490. eCollection 2014. PMID 24904503
- [Background] Tenenbaum EJ, Sobel DM, Sheinkopf SJ, Shah RJ, Malle BF, Morgan JL. Attention to the mouth and gaze following in infancy predict language development. J Child Lang. 2015 Nov;42(6):1173-90. doi: 10.1017/S0305000914000725. Epub 2014 Nov 18. PMID 25403090
- [Background] Lewkowicz DJ, Hansen-Tift AM. Infants deploy selective attention to the mouth of a talking face when learning speech. Proc Natl Acad Sci U S A. 2012 Jan 31;109(5):1431-6. doi: 10.1073/pnas.1114783109. Epub 2012 Jan 17. PMID 22307596
- [Background] Tenenbaum EJ, Shah RJ, Sobel DM, Malle BF, Morgan JL. Increased focus on the mouth among infants in the first year of life: A longitudinal eye-tracking study. Infancy. 2013 Jul;18(4):534-553. doi: 10.1111/j.1532-7078.2012.00135.x. PMID 23869196
- [Background] Bottema-Beutel K, Yoder PJ, Hochman JM, Watson LR. The role of supported joint engagement and parent utterances in language and social communication development in children with autism spectrum disorder. J Autism Dev Disord. 2014 Sep;44(9):2162-74. doi: 10.1007/s10803-014-2092-z. PMID 24658867